CLINICAL TRIAL: NCT01977690
Title: Clavicle Splint for Pain Reduction After Posterior Cervicothoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stephan Duetzmann, M.D.,M.Sc., Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLABRA
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Posterior Cervical Surgery; Posterior Cervical Fusion; Posterior Cervical Laminectomy; Posterior Cervical Laminoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Management (No Intervention): Patients wore no brace.
- Clavicle Brace Wearing (Experimental): Patient has to wear clavicle brace for one month.
  Interventions: Device: Clavicle Brace

INTERVENTIONS:
Device: Clavicle Brace
  Arms: Clavicle Brace Wearing

SUMMARY:
The purpose of the study is to see whether a clavicle splint can decrease the pain after posterior cervicothoracic surgery. The term "cervicle splint" conveys that the investigators do not deal with clavicle fractures here but use the splint he stabilize the posterior cervical area. The investigators want to demonstrate this in a prospective randomized manner.

DETAILED DESCRIPTION:
In this prospectively controlled randomized study 30 patients who had undergone posterior cervical spine surgery were randomized into two groups who either wore or did not wear a clavicle brace to retract the shoulders. Patients in the brace group began wearing the brace on postoperative day 4, and continuously wore it throughout the 30-day study period. Outcome was measured as daily levels of self-reported pain and number of pain pills taken during the 30-day postoperative period. .

After hypothesizing a mean pain reduction through the brace on the visual analog scale (VAS) for pain from 5 to 3 with a standard deviation of 1, we calculated that at a power level of 99% and an alpha error of 5%, and given that the VAS numbers were normally distributed, we needed 22 patients to enroll into the study. We increased this number to 30 to account for early and late dropouts.

The study was performed at a single institution with patients from 2 different spine surgeons.

Patients were randomized prior to or the day after the procedure to either wear or not wear the clavicle brace. Randomization was done through closed envelopes that the patients drew. Dissection was performed by the two fellows at our institution and depended solely on the number of fused levels and whether or not a tumor had to be removed. Closure was also performed by the two spine fellows after instruction by the senior author. Cervical alignment was reviewed using the C2-C7 angle according to Cobb's method on lateral images. The cervico-thoracic angles were calculated by the addition of the cervical spine angle and the remaining angles of thoracic spine until T3 according to Cobb's method.

The brace was provided by the hospital. Patients were instructed how to properly wear the brace by the first author, the senior author, or the hospital Rehabilitation Orthotics specialist. To complete the study, patients wore the brace for at least 30 days. (Patients of J.P. continued to wear the brace for 3 months outside of the study period.). All patients wore hard cervical collars until the end of the study period.

Patients self-recorded their average level of pain on a scale from 1 to 10 for each post-surgery day beginning on postoperative day 2. They also recorded the number of pain pills they took each day. On the same sheet used to record medication usage, patients were instructed to record each day whether they were able to wear the brace or if they experienced problems. At their 1 month postoperative visit the incision was inspected and palpated by the first or senior author for the presence of fascial dehiscence and its occurrence was recorded.

Every patient routinely received narcotic and non-narcotic pain medication on an as-needed basis in the hospital. No nonsteroidal anti-inflammatory drugs, such as ibuprofen or ketorolac, were given. If, on a particular postoperative day, patients were still on an intravenous narcotic patient-controlled anesthesia (PCA), that day's data were not recorded for the study.

ELIGIBILITY:
Inclusion Criteria:

- Patient underwent cervicothoracic surgery from posterior -

Exclusion Criteria:

- Patients that are potentially vulnerable

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Duetzmann, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duetzmann S, Cole T, Senft C, Seifert V, Ratliff JK, Park J. Clavicle pain and reduction of incisional and fascial pain after posterior cervical surgery. J Neurosurg Spine. 2015 Dec;23(6):684-9. doi: 10.3171/2015.2.SPINE141118. Epub 2015 Aug 21. PMID 26296190

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Management: Patients received analgesics ad libitum
- Clavicle Brace Wearing: Patient has to wear clavicle brace for one month.
  Clavicle Brace
Period: Overall Study
Arm/Group | Standard Management | Clavicle Brace Wearing
Started | 15 | 15
Completed | 15 | 11
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Standard Management: Every patient routinely received narcotic and non-narcotic pain medication on an as-needed basis in the hospital. No nonsteroidal anti-inflammatory drugs, such as ibuprofen or ketorolac, were given.
- Total: Total of all reporting groups
Arm/Group | Standard Management | Clavicle Brace Wearing | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 55 [41 to 79] | 57 [45 to 84] | 56 [41 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Average Neck Pain Level
Description: Patients self-recorded their average level of pain on a scale from 1 to 10 for each post-surgery day beginning on postoperative day 2. 1 Meaning least pain, 10 meaning worst level of pain
Time Frame: 1 month
Population: 4 participants in the Clavicle brace group did not tolerate the brace and are included in the standard management group for this analysis. Only participants will available data are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale (VAS pain scale)
Arm/Group | Standard Management | Clavicle Brace Wearing
Number analyzed (Participants) | 16 | 11
units on a scale (VAS pain scale) | 1 (1) | 1 (1)

ADVERSE EVENTS:
Description: Adverse events are reported according to randomization group.
Groups:
- Standard Management: Patients received analgesic ad libitum
Arm/Group | Standard Management | Clavicle Brace Wearing
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Small number of patients and its location at a single institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes